CLINICAL TRIAL: NCT02176577
Title: An Open-Label, Multi-Center Study to Determine the Pharmacokinetics of Product 0405 in the Treatment of Atopic Dermatitis in Adolescent Subjects
Brief Title: Study to Determine the Pharmacokinetics of Product 0405
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0405-01-07
Record Dates: First submitted 2014-06-17; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Product 0405 (Experimental): Topically Active Investigational Product 0405
  Interventions: Drug: Product 0405

INTERVENTIONS:
Drug: Product 0405 — Product 0405 will be administered topically, twice daily for 28 days.

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics of Product 0405 in the Treatment of Atopic Dermatitis in Adolescent Subjects.

DETAILED DESCRIPTION:
Treament medication will be administered topically twice daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis
* Good health with the exception of Atopic Dermatitis
* Percent body surface area minimums

Exclusion Criteria:

* Subject who are nursing, pregnant or planning a pregnancy

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Phamacokinetic sampling | 28 days

SECONDARY OUTCOMES:
Laboratory tests, vital signs, adverse events and local skin safety signs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Kaplan, Study Director — Fougera Pharmaceuticals Inc.